CLINICAL TRIAL: NCT00321698
Title: Phase I/II Study of Preoperative Radiation and Docetaxel Activity in High Risk Localized Prostate Cancer
Brief Title: Radiation Therapy and Docetaxel in Treating Patients Who Are Undergoing Surgery for Localized Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding withdrawal
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Principal Investigator, Mark Garzotto, MD, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00001581; IIT16179 (Other Grant/Funding Number: Sanofi-Aventis funding number); OHSU-1581 (Other: OHSU IRB number); PVAMC-11-1205/ M1675 (Other: Portland VA IRB numbers); OHSU-SOL-05077-L (Other: OHSU Knight Cancer Institute number); CDR0000467219 (Other: NCI PDQ ID); NCI-2012-01122 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Results first posted 2016-12-30 (Estimated); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage II prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Radiotherapy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase I Dose 1-4 (Experimental): Group 1=radiation only; Group 2=Docetaxel IV over 30mins, 10mg/m2; weekly x 5 weeks starting on day one of radiation; Group 3=Docetaxel IV over 30mins, 20mg/m2; weekly x 5 weeks starting on day one of radiation; Group 4=Docetaxel IV over 30mins, 30mg/m2; weekly x 5 weeks starting on day one of radiation
  Radiation: All men receive same radiation treatment protocol. External Beam, 45 Gy (1.8 Gy fractions), 5 per week (daily) x 5 weeks (25 fractions)
  Interventions: Radiation: Intensity-Modulated Radiation Therapy (IMRT); Drug: Docetaxel+IMRT
- Phase II MTD Dose (Experimental): Phase II with no phase I dose-limiting toxicities=Docetaxel IV over 30mins, 30mg/m2; weekly x 5 weeks starting on day one of radiation
  Radiation: All men receive same radiation treatment protocol. External Beam, 45 Gy (1.8 Gy fractions), 5 per week (daily) x 5 weeks (25 fractions)
  Interventions: Drug: Docetaxel+IMRT

INTERVENTIONS:
Radiation: Intensity-Modulated Radiation Therapy (IMRT) — Group 1=radiation only; All men in all Arms/Groups receive same radiation treatment protocol. External Beam, 45 Gy (1.8 Gy fractions), 5 per week (daily) x 5 weeks (25 fractions)
  Other Names: Radiation therapy
  Arms: Phase I Dose 1-4
Drug: Docetaxel+IMRT — Group 2=IV over 30mins, 10mg/m2; weekly x 5 weeks starting on day one of radiation; Group 3=IV over 30mins, 20mg/m2; weekly x 5 weeks starting on day one of radiation; Group 4=IV over 30mins, 30mg/m2; weekly x 5 weeks starting on day one of radiation; Phase II with no phase I dose-limiting toxicities=IV over 30mins, 30mg/m2; weekly x 5 weeks starting on day one of radiation
  Radiation: All men receive same radiation treatment protocol. External Beam, 45 Gy (1.8 Gy fractions), 5 per week (daily) x 5 weeks (25 fractions)
  Other Names: Chemotherapy with Radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy together with chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase I/II trial is studying the side effects and best dose of docetaxel when given together with radiation therapy and to see how well they work in treating patients who are undergoing surgery for high-risk localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) of neoadjuvant radiotherapy and docetaxel in patients who are undergoing prostatectomy for high-risk localized prostate cancer.
* Determine the pathologic response rate in patients treated at the phase II dose.

Secondary

* Determine the prostate-specific antigen (PSA) short-term response rate in patients treated with this regimen.
* Determine the long-term safety of this regimen prior to radical prostatectomy in these patients.
* Determine the clinical response to this regimen by urologic examination of these patients.
* Determine the surgical margin status at the time of prostatectomy in patients treated with this regimen.
* Determine the effect of this regimen, in terms of Health-Related Quality of Life by Expanded Prostate Cancer Index Composite (EPIC) and urinary symptom scores by the American Urological Association's measures, in these patients.
* Determine the clinical progression-free rate in patients treated with this regimen.
* Identify pretreatment predictors of response in these patients by examining tissue biomarkers in preserved pretreatment biopsy specimens.
* Determine the biologic impact of this regimen on these patients by examining the prostatectomy specimens.
* Collect frozen serum for future analysis of correlative biomarkers.
* Compare the RNA content (gene expression profile) of pre- and post-treatment tumor specimens in order to describe the molecular impact of this regimen on prostate cancer.

OUTLINE: This is a phase I, dose-escalation study of docetaxel followed by a phase II study. All patients undergo a biopsy of the prostate to gather research-only specimens prior to the beginning of treatment.

* Phase I: Patients undergo radiotherapy once daily, 5 days a week, for 5 weeks. Patients also receive docetaxel IV on days 1, 8, 15, 22, and 29. Treatment continues in the absence of disease progression or unacceptable toxicity. Approximately 4-6 weeks after completion of chemoradiotherapy, patients undergo a radical prostatectomy.

Cohorts of 3-6 patients receive escalating doses of docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience a dose-limiting toxicity. At least 6 patients are treated at the MTD.

* Phase II: Patients undergo radiotherapy as in phase I. Patients also receive docetaxel at the MTD determined in phase I and then undergo prostatectomy as in phase I.

PROJECTED ACCRUAL: A total of 42 patients will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA; DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Localized disease, meeting 1 of the following staging criteria:

    * Clinical stage T2b (palpable bilateral movement) disease
    * Surgically resectable T3 disease
* Meets any of the following high-risk* features:

  * PSA ≥ 15 ng/mL
  * Gleason grade ≥ 4+3 (4+3, 4+4, or 5+any, but not 3+4) NOTE: *High risk defined as > 50% chance of failure with local therapy
* Plans to undergo prostatectomy as primary therapy
* No evidence of lymph nodes ≥ 2 cm in diameter by pelvic CT scan

  * Scan only required in patients with a PSA ≥ 40 ng/mL
* No evidence of bone metastases by bone scan

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 10 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* White blood cell (WBC) > 3,000/mm^3
* Neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Direct bilirubin normal
* Alanine aminotransferase (ALT) < 2.0 times upper limit of normal (ULN) (1.5 times ULN if alkaline phosphatase [AP] > 2.5 times ULN)
* Alkaline phosphatase (AP) < 4.0 times ULN
* No other serious medical condition that would preclude study treatment
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* No peripheral neuropathy ≥ grade 2
* No hypersensitivity to drugs formulated with polysorbate 80
* No significant contraindications to corticosteroids
* No history of scleroderma
* No active inflammatory bowel disease (IBD) or IBD that is being medically treated

  * Inclusion of patients with a remote history of IBD is at the discretion of radiotherapist

EXCLUSION CRITERIA; PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior therapy for prostate cancer, including any of the following:

  * Conventional hormonal therapy (e.g., orchiectomy, luteinizing hormone-releasing hormone therapy, antiandrogen therapy, or estrogen therapy)
  * External-beam radiotherapy or brachytherapy
  * Cryotherapy
  * Cytotoxic chemotherapy
* No prior pelvic radiotherapy

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-04-21 (Actual); Primary Completion 2009-10-01 (Actual); Study Completion 2023-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Garzotto, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - OHSU Knight Cancer Institute, Portland, Oregon

REFERENCES:
- [Derived] Ohaegbulam KC, Post CM, Farris PE, Garzotto M, Beer TM, Hung A, Williamson CW. Safety and Efficacy of Neoadjuvant Docetaxel and Radiotherapy in Localized High-Risk Prostate Cancer: Results From a Prospective Pilot Study. Am J Clin Oncol. 2025 Feb 1;48(2):75-82. doi: 10.1097/COC.0000000000001151. Epub 2024 Oct 30. PMID 39473059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject accrual from Urology clinics started in April 2006; annual follow-up of 22 VA, 3 Oregon Health & Science University (OHSU) (25 total) subjects who completed ended in 2011; 10 year follow-up of these patients will be completed in 2021.
Pre-assignment Details: Our 1 screen failure was excluded as a result of having a different type of cancer, other than non-melanoma skin cancer, within the past 5 years.
Groups:
- Phase I, Radiation Only: Group 1=radiation only;
  Radiation: All men receive same radiation treatment protocol. External Beam, 45 Gy (1.8 Gy fractions), 5 per week (daily) x 5 weeks (25 fractions)
- Phase I, Dose 1: Group 2=IV over 30mins, 10mg/m2 weekly x 5 weeks starting on day one of radiation;
  Radiation: All men receive same radiation treatment protocol. External Beam, 45 Gy (1.8 Gy fractions), 5 per week (daily) x 5 weeks (25 fractions)
  Chemotherapy (Groups 2-4): Docetaxel IV over 30mins weekly x 5 weeks starting on day one of radiation. The maximum planned dose of 30 mg/m2 was reached without Dose-Limiting Toxicities.
- Phase I, Dose 2: Group 3=IV over 30mins, 20mg/m2 weekly x 5 weeks starting on day one of radiation;
  Radiation: All men receive same radiation treatment protocol. External Beam, 45 Gy (1.8 Gy fractions), 5 per week (daily) x 5 weeks (25 fractions)
  Chemotherapy (Groups 2-4): Docetaxel IV over 30mins weekly x 5 weeks starting on day one of radiation. The maximum planned dose of 30 mg/m2 was reached without Dose-Limiting Toxicities.
- Phase I, Dose 3: Group 4=IV over 30mins, 30mg/m2 weekly x 5 weeks starting on day one of radiation;
  Radiation: All men receive same radiation treatment protocol. External Beam, 45 Gy (1.8 Gy fractions), 5 per week (daily) x 5 weeks (25 fractions)
  Chemotherapy (Groups 2-4): Docetaxel IV over 30mins weekly x 5 weeks starting on day one of radiation. The maximum planned dose of 30 mg/m2 was reached without Dose-Limiting Toxicities.
- Phase II, MTD Dose: MTD=Docetaxel IV over 30mins, 30mg/m2 weekly x 5 weeks starting on day one of radiation plus external beam radiation, 45 Gy (1.8 Gy fractions), 5 per week (daily) x 5 weeks (25 fractions).
  Radiation: All men receive same radiation treatment protocol. External Beam, 45 Gy (1.8 Gy fractions), 5 per week (daily) x 5 weeks (25 fractions)
Period: Phase I, Rad Only & Dose 1-3
Arm/Group | Phase I, Radiation Only | Phase I, Dose 1 | Phase I, Dose 2 | Phase I, Dose 3 | Phase II, MTD Dose
Started | 3 | 3 | 3 | 3 | 0
Completed | 3 | 3 | 3 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Phase II, MTD Dose
Arm/Group | Phase I, Radiation Only | Phase I, Dose 1 | Phase I, Dose 2 | Phase I, Dose 3 | Phase II, MTD Dose
Started | 0 | 0 | 0 | 0 | 13 (+1 screen failure)
Completed | 0 | 0 | 0 | 0 | 13
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I, Radiation Only: Drug: N/A
  4 groups of men in phase I study.
  Group 1=radiation only
  Radiation: radiation therapy
  All men receive same radiation treatment protocol. External Beam, 45 Gy (1.8 Gy fractions), 5 per week (daily) x 5 weeks (25 fractions)
- Phase I, Dose 1: Drug: docetaxel
  4 groups of men in phase I study.
  Group 2=IV over 30mins, 10mg/m2; weekly x 5 weeks starting on day one of radiation;
  Radiation: radiation therapy
  All men receive same radiation treatment protocol. External Beam, 45 Gy (1.8 Gy fractions), 5 per week (daily) x 5 weeks (25 fractions)
- Phase I, Dose 2: Drug: docetaxel
  4 groups of men in phase I study.
  Group 3=IV over 30mins, 20mg/m2; weekly x 5 weeks starting on day one of radiation;
  Radiation: radiation therapy
  All men receive same radiation treatment protocol. External Beam, 45 Gy (1.8 Gy fractions), 5 per week (daily) x 5 weeks (25 fractions)
- Phase I, Dose 3: Drug: docetaxel
  4 groups of men in phase I study.
  Group 4=IV over 30mins, 30mg/m2; weekly x 5 weeks starting on day one of radiation
  Radiation: radiation therapy
  All men receive same radiation treatment protocol. External Beam, 45 Gy (1.8 Gy fractions), 5 per week (daily) x 5 weeks (25 fractions)
- Phase II, MTD Dose: Drug: docetaxel
  Phase II with no phase I dose-limiting toxicities=IV over 30mins, 30mg/m2; weekly x 5 weeks starting on day one of radiation
  Radiation: radiation therapy
  All men receive same radiation treatment protocol. External Beam, 45 Gy (1.8 Gy fractions), 5 per week (daily) x 5 weeks (25 fractions)
- Total: Total of all reporting groups
Arm/Group | Phase I, Radiation Only | Phase I, Dose 1 | Phase I, Dose 2 | Phase I, Dose 3 | Phase II, MTD Dose | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 2 | 3 | 11 | 20
  >=65 years | 1 | 1 | 1 | 0 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.67 (8.14) | 62.67 (7.64) | 66.33 (4.93) | 58.00 (6.56) | 60.54 (4.58) | 61.92 (5.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 3 | 13 | 25
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: Maximal tolerated dose (MTD) of the combination radiation (45 Gy) and docetaxel.
  The dose of radiation will be fixed at 45 Gy while the dose of docetaxel will be escalated. The starting dose of docetaxel will be 10 mg/m2 and will be escalated in increments of 10 mg/m2 up to a dose of 30 mg/m2 the pre-planned ceiling).
  MTD will be the dose that is associated with no more than 1 dose limiting toxicity (DLT) up to 6 patients. The DLT will be defined as clinically significant grade 3 non-hematologic or grade 4 hematologic toxicity, attributable to the chemoirradiation. If 2 of 3 patients experience a DLT, dose escalation will stop and the previous dose level will be considered the MTD. If 1 of 3 has DLT, additional 3 patients will be enrolled at the same dose level. If none of the additional 3 patients has DLT, the dose escalation will continue. If 1 additional patient has DLT, the previous dose will be considered the MTD and dose escalation will be stopped.
Time Frame: 5 weeks
Population: Outcome analysis includes the subjects from all 4 phase I groups, inclusive of subjects who only received radiation, as all subjects across all phases received the same radiation dosage. Phase I, group 1 subjects were included in case MTD was zero.
Measure: Number; unit: mg/m^2
Groups:
- Phase I Dose 1-4: 4 groups of men in phase I study.
  Group 1=radiation only; Group 2=IV over 30mins, 10mg/m2; weekly x 5 weeks starting on day one of radiation; Group 3=IV over 30mins, 20mg/m2; weekly x 5 weeks starting on day one of radiation; Group 4=IV over 30mins, 30mg/m2; weekly x 5 weeks starting on day one of radiation.
Arm/Group | Phase I Dose 1-4
Number analyzed (Participants) | 12
mg/m^2 | 30

2. Primary Outcome: Pathologic Response Rate at the Phase II Dose
Description: Pathologic response rate is determined post-prostatectomy by pathologist laboratory analyses. The TNM system is the most widely used cancer staging system. Most hospitals and medical centers use the TNM system as their main method for cancer reporting. In the TNM system:
  The T refers to the size and extent of the main/primary tumor. T1, T2, T3, T4: Refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail, such as T3a and T3b.
Time Frame: 4-6 weeks after study treatment
Measure: Number; unit: participants
Arm/Group | Phase II MTD Dose
Number analyzed (Participants) | 13
participants
  Pathologic Stage pT2c | 7
  Pathologic Stage pT3a | 3
  Pathologic Stage pT3b | 3

3. Secondary Outcome: Prostate-specific Antigen Short-term Response Rate Measured as a Percentage Change in PSA
Description: All participants were combined for this assessment as pre-specified in the protocol.
  The percentage change for patients were determined from pre- and post- treatment PSA values. The mean percentage change in PSA will be reported.
  PSA will be monitored every 3-6 months during the first 5 years, then annually after surgery for up to 10 years
Time Frame: Baseline (pre-treatment) and 1 month after surgery (post-treatment)
Population: Pre- and post-treatment PSA values were available in 22 of 25 patients.
Measure: Mean (95% Confidence Interval); unit: percentage change
Groups:
- All Research Participants: This Outcome Measure was assessed in aggregate, combining participants from both phases of the study, as per the planned protocol.
  Phase I: Group 1=radiation only; Group 2=IV over 30mins, 10mg/m2; weekly x 5 weeks starting on day one of radiation; Group 3=IV over 30mins, 20mg/m2; weekly x 5 weeks starting on day one of radiation; Group 4=IV over 30mins, 30mg/m2; weekly x 5 weeks starting on day one of radiation.
  Phase II: Phase II with no phase I dose-limiting toxicities=Docetaxel IV over 30mins, 30mg/m2; weekly x 5 weeks starting on day one of radiation.
  Radiation: All men receive same radiation treatment protocol. External Beam, 45 Gy (1.8 Gy fractions), 5 per week (daily) x 5 weeks (25 fractions).
Arm/Group | All Research Participants
Number analyzed (Participants) | 22
percentage change | -49.1 [-60.3 to -36.7]

4. Secondary Outcome: Long-term Safety
Description: An adverse event is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure.
Time Frame: Regular intervals both study-related and clinical standard of care-related; assessed at end of study treatment. Average timeframe to follow safety was 1 year and includes all grade 3-4 adverse events
Population: Phase I participants numbered 12 (receiving different chemotherapy doses) and Phase II participants numbered 13 (receiving the maximally tolerated chemotherapy dose). This Outcome Measure was assessed in aggregate, combining participants from both phases of the study, per protocol.
Measure: Number; unit: grade 3-4 adverse events
Arm/Group | Phase I Dose 1-4 | Phase II MTD Dose
Number analyzed (Participants) | 12 | 13
grade 3-4 adverse events | 9 | 8

5. Secondary Outcome: Clinical Response to Treatment as Measured by Urologic Examination
Description: Biochemical Recurrence is defined as a detectable or rising PSA value after surgery that is 0.2 ng/mL or greater with a second confirmatory level of 0.2 ng/mL or greater.
Time Frame: Each participant was examined 3, 6, 9, 12 months, and annually for an average of 10 years after surgery.
Population: Clinical response to treatment was measured by regular Prostatic Specific Antigen (PSA) blood draws. The following men per chemotherapy dosage experienced a detectable or rising PSA value after surgery with a 2nd confirmatory level of 0.2ng/mL or higher (defined as biochemical recurrence of prostate cancer).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I, Radiation Only | Phase I, Dose 1 | Phase I, Dose 2 | Phase I, Dose 3 | Phase II, MTD Dose
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 13
Participants | 1 | 2 | 0 | 2 | 5

6. Secondary Outcome: Surgical Margin Status at Time of Prostatectomy (Count of Subjects With Negative Surgical Margins)
Description: Pathologic response rate is determined post-prostatectomy by pathologist laboratory analyses. The TNM system is the most widely used cancer staging system. Most hospitals and medical centers use the TNM system as their main method for cancer reporting. In the TNM system:
  The M refers to whether the cancer has metastasized. This means that the cancer has spread outside of the primary tumor to other parts of the body.
Time Frame: 5 weeks
Population: For Phase I Dose 1-4, all participants were combined for this assessment as pre-specified in the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose 1-4 | Phase II MTD Dose
Number analyzed (Participants) | 12 | 13
Participants | 9 | 13

7. Secondary Outcome: Efficacy Assessed Using Health-Related Quality of Life by Expanded Prostate Cancer Index Composite and Urinary Symptom Scores by American Urological Association's Measures
Description: Mean change in score from Baseline to 12-months pot-op. A single outcome, Health Related Quality of Life (QOL), was specified in the protocol. All 6 score means and confidence intervals are reported here as a single outcome; a separate row for each score.
  AUA Symptom Score is designed to measure lower urinary tract symptoms (LUTS) resulting from benign prostatic hyperplasia or other causes in men. Higher scores indicate more LUTS (scale 0-35). 1-7, mild; 8-19, moderate; 20-35, severe.
  EPIC quality of life instruments is a 32-item self-report questionnaire that measures the QOL of prostate cancer patients. 4 subscales measuring urinary (further consisting of two sub-components, EPIC Urinary Incontinence Score and EPIC Urinary Obstructive/Irritative Score), bowel, sexual and hormonal changes. Scores for each of the subscales, as well as for each sub-component within the Urinary sub scale, are transformed linearly to a 0-100 scale with higher scores representing better QOL.
Time Frame: Baseline and 12 Months Post-Prostatectomy
Population: Scores not available for some participants
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | All Research Participants
Number analyzed (Participants) | 25
units on a scale
  AUA Symptom Score: number analyzed (Participants) | 24
  AUA Symptom Score | 0.67 [-2.96 to 4.29]
  EPIC Urinary Incontinence Score: number analyzed (Participants) | 21
  EPIC Urinary Incontinence Score | -36.52 [-51.38 to -21.67]
  EPIC Urinary Obstructive/Irritative Score: number analyzed (Participants) | 22
  EPIC Urinary Obstructive/Irritative Score | 3.41 [-5.55 to 12.37]
  EPIC Bowel | 1.45 [-6.42 to 9.33]
  EPIC Hormonal: number analyzed (Participants) | 23
  EPIC Hormonal | 0.00 [-6.42 to 6.42]
  EPIC Sexual: number analyzed (Participants) | 22
  EPIC Sexual | -36.26 [-48.84 to -23.68]

8. Secondary Outcome: Clinical Progression-free Rate as Determined by <0.1ng PSA Results
Description: The estimated percentage of participants who were progression-free at 5 years per analyses of PSA results post-study treatment.
Time Frame: 3, 6, 9, 12 months and annually, up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Research Participants
Number analyzed (Participants) | 25
percentage of participants | 62.8 [41.9 to 83.6]

ADVERSE EVENTS:
Time Frame: Timeframe to follow safety was up to 1 year, for an average of 133.84 days per subject.
Description: For each subject, adverse events (AEs) are reported from the time of trial entry to 6 weeks post-surgery.
  Serious adverse events (SAEs) (grade 3-4) are all related to treatment. Only Serious grade 3 and higher AEs related to treatment were recorded as specified per protocol.
Arm/Group | Phase I, Radiation Only | Phase I, Dose 1 | Phase I, Dose 2 | Phase I, Dose 3 | Phase II, MTD Dose
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/3 | 3/3 | 3/3 | 8/13
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Radiation Only (N=3) | Phase I, Dose 1 (N=3) | Phase I, Dose 2 (N=3) | Phase I, Dose 3 (N=3) | Phase II, MTD Dose (N=13)
Difficulty with ADLs (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) — Difficulty with activities of daily living (ADLs)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Lymphapenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 5 (5)
Hemoglobin (L) (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Patient accrual was not completed due to the sponsor withdrawing funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No